CLINICAL TRIAL: NCT06659952
Title: A Prospective Study of HIV+ Deceased Donor Heart Transplant for HIV+ Recipients
Brief Title: HIV+ Deceased Donor Heart Transplant Study for HIV+ Recipients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ricardo La Hoz, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2024-0777
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: HIV Infection; Advanced End Stage Heart Failure
Keywords: HIV positive donor; HIV positive recipient; Heart transplant
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: "Natural randomization" will take place as OPTN organ offers become available and will be assigned to either arm based on whether the subject accepts/ declines the HIV+ donor heart.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV D+/R+ Arm (Experimental): If HIV+ donor heart is available prior to HIV-negative donor heart, HIV-positive participant who agreed to receive HIV+ donor heart as part of this study receives the organ (heart) from an HIV- positive donor.
  Interventions: Other: HIV-positive heart transplant
- HIV D-/R+ Arm (Control Arm) (No Intervention): If HIV- donor heart is available first, the HIV-positive participant receives the organ (heart) from an HIV- negative donor as part of standard organ waitlist/ clinical care.

INTERVENTIONS:
Other: HIV-positive heart transplant — Receipt of heart from HIV-positive deceased donor only as part of this study
  Arms: HIV D+/R+ Arm

SUMMARY:
This will be a prospective single-center interventional trial to compare the outcomes of HIV-positive heart transplant recipients by the HIV status of the donor; HIV-positive vs. HIV-negative and learn whether heart organ transplantation from HIV+ deceased donors is as safe and effective in HIV+ recipients as transplants from HIV- deceased donors.

Patient will undergo standard evaluation for eligibility of transplantation by the primary heart transplant team. If patient meets eligibility criteria, they will be informed about the study and consent will be obtained. Informed consent will be obtained in a private clinic or inpatient hospital room in a confidential setting. HIV-positive or HIV-negative offers will be made by Organ Procurement and Transplantation Network (OPTN) (serving as a means of "natural randomization" and this information will also be collected, along with the information regarding any information for primary offer declines from the patients as well as other clinical indications to decline an organ offer. As a result of this, there will be two main groups in the study participants that will undergo analysis:

1. patients/recipients that are HIV+ who receive an organ from an HIV+ donor (HIV D+/R+ group)
2. patients/recipients that are HIV+ who receive an organ from an HIV negative donor (HIV D-/R+ group)

Only study participants will be able to receive organ offers from both HIV-positive and HIV-negative organ donors whichever is available first regardless of HIV status. This is the only study intervention. Baseline visit parameters will be obtained during a routine heart transplant visit. There will be no additional procedures or blood collection after the baseline study visit.

Study data will be collected from chart review of routine post-transplant follow-up visits at weeks 52 (1 year), 104 (2 years), and 152 (3 years) after the transplant.

DETAILED DESCRIPTION:
The primary objective is to evaluate the safety of heart transplantation in HIV-positive recipients and to study any potential complications of solid organ transplantation in the recipient, as well as assess the long-term health and mortality.

Secondary objectives are to compare other clinical outcomes between HIV+ transplant recipients of hearts from HIV+ and HIV- donors.

HIV D+/R+ transplantation is still less common than HIV D-/R+ transplantation due to the overall availability of donor organs. Additionally, most of the HIV D+/R+ transplants have been done for kidney transplants. Overall, there is more data accruing regarding transplantation and HIV disease, but most of the procedures are done in the kidney and liver organ systems. Not only is it important to further expand the donor pool for patients with HIV and heart failure, further data is needed in thoracic organ transplantation and HIV-positive recipients. The HIV Organ Policy Equity Act (HOPE Act - enacted on November 21, 2013), made it possible for an HIV+ recipient to receive an HIV+ organ as a part of a research study.

HIV+ Deceased Donor Criteria:

1. Donation after brain death or cardiac death.
2. HIV+ donors have confirmed or suspected HIV infection* (by medical record history and/or a licensed HIV test.) If HIV infection is diagnosed during the donor evaluation process, a second confirmatory test will be required).
3. Donor has no active opportunistic infections, neoplasms, or severe acute retroviral syndrome; if previous history of an opportunistic infection, donor has received appropriate treatment.
4. Donors may have any HIV-1 RNA viral load provided a safe, tolerable and effective post-transplant antiretroviral regimen to be prescribed for the recipient is anticipated, described and justified.
5. Donors with active hepatitis C virus (HCV) infection (detectable HCV nucleic acid by licensed assay in a Clinical Laboratory Improvement Amendments (CLIA) certified lab are acceptable based on local site practice.

ELIGIBILITY:
Inclusion Criteria:

All individuals with advanced heart failure and HIV infection who meet the study inclusion and exclusion criteria will be eligible for participation in the study.

* Participant meets the standard criteria for heart transplant at the local center.
* Participant is able to understand and provide informed consent.
* Participant meets with an independent advocate per the HOPE Act Safeguards and Research Criteria.
* Documented HIV infection (by any licensed assay, or documented history of detectable HIV-1 RNA).*
* Participant is ≥ 18 years old.
* Opportunistic complications: if prior history of an opportunistic infection, the participant has received appropriate therapy and has no evidence of active disease. Medical record documentation should be provided whenever possible.*
* CD4+ (cluster of differentiation 4+) T-cell count: ≥ 200/μL within 16 weeks of transplant.*
* HIV-1 RNA is below 50 copies RNA/mL.*/** Viral blips between 50-400 copies will be allowed as long as there are not consecutive measurements > 200 copies/mL. **Organ recipients who are unable to tolerate ART due to organ failure or recently started Antiretroviral Therapy (ART) may have detectable viral load and still be eligible if a safe and effective antiretroviral regimen to be used by the recipient after transplantation is described.
* Participant is willing to comply with all medications related to their transplant and HIV management.
* For participants with a history of aspergillus colonization or disease, no evidence of active disease.
* The participant must have or be willing to start seeing a primary medical care provider with expertise in HIV management.
* Agreement to use contraception; according to the FDA Office of Women's Health (http://www.fda.gov/birthcontrol), there are a number of birth control methods that are more than 80% effective. Female participants of child-bearing potential must consult with their physician and determine the most suitable method(s) from this list to be used from the time that study treatment begins until after study completion.
* Participant is not suffering from significant wasting (e.g. body mass index < 21) thought to be related to HIV disease.

Exclusion Criteria:

Individuals who meet any of these criteria are not eligible for enrollment as study participants:

* Participant has a history of progressive multifocal leukoencephalopathy (PML) or primary central nervous system (CNS) lymphoma.*
* Participant is pregnant or breastfeeding. (Note: Participants who become pregnant post-transplant will continue to be followed in the study and will be managed per local site practice. Women that become pregnant should not breastfeed.)
* Past or current medical problems or findings from medical history, physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2034-10 (Estimated); Study Completion 2034-10 (Estimated)

PRIMARY OUTCOMES:
Time to a composite event of all-cause-mortality, graft failure, graft function | 4 years post-transplant
  Time to event outcome measured as the time from randomization to the occurrence of the first event.

SECONDARY OUTCOMES:
Number of participants who survived | 4 years post-transplant
  Count of participants who survived
Incidence of Graft survival | 4 years post-transplant
  Graft survival: Survival without re-transplantation or death related to graft dysfunction
Number of Participants With One or More Serious Adverse Experience (SAE) | 4 years post-transplant
  Count of Participants With One or More Serious Adverse Experience (SAE) post transplant is assessed
Number of participants with graft rejection | 4 years post-transplant
  Count of participants with graft rejection will be reported. Rejections will be defined by pathologist and clinician.
Incidence of graft function | 4 years post-transplant
  Graft function will be assessed by echocardiography - Left Ventricular ejection function

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo La Hoz, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No